CLINICAL TRIAL: NCT04197635
Title: Short-term Effects of Dapagliflozin on Peak VO2 in Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: Short-term Effects of Dapagliflozin on Peak VO2 in HFrEF
Acronym: DAPA-VO2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Julio Nuñez, Principal Investigator, Clinical Professor, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-17-13447(DAPA-HF); 2018-002614-12 (EudraCT Number)
Record Dates: First submitted 2019-11-01; First posted 2019-12-13 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure with Reduced Ejection Fraction; Functional Capacity; Quality of life
MeSH Terms: interventions — Echocardiography; Diastole; Quality of Life; Walk Test

STUDY DESIGN:
Intervention Model Description: This study will be a double-blind multicenter randomized study (1:1) to evaluate the effect of dapagliflozin 10 mg per day or placebo on short-term functional capacity evaluated through changes in peak oxygen consumption The patients will be randomized to receive dapagliflozin or placebo. Once the inclusion criteria are fulfilled and the informed consent signed, patients will be randomized, and efficacy endpoints will be evaluated at 3 time points: 1) baseline (before dapagliflozin/placebo administration), 2) 30 days after randomization, and, 3) 90 days after randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After providing informed consent, patients will be randomly assigned, with a remote, web-based computer-generated block randomization procedure in an allocation 1:1 ratio, to either receive dapagliflozin 10 mg per day or placebo (one tablet a day orally). This system will allow the maintenance of the randomization codes and the opening of them if necessary. Investigators and patients will be blinded to treatment allocations.
  Knowing that no treatment crossings between both groups are expected, there is no need of planning washing periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10 mg (Active Comparator): After providing informed consent, patients will be randomly assigned to receive dapagliflozin 10 mg per day.
  Interventions: Diagnostic Test: Maximal functional capacity by cardiopulmonary exercise testing; Diagnostic Test: Echocardiography; Behavioral: Evaluation of health related quality of life; Diagnostic Test: Submáximal functional capacity assesment by 6 minutes walk test; Other: Clinical evaluation
- Placebo identical to dapagliflozin 10 mg (Placebo Comparator): After providing informed consent, patients will be randomly assigned to receive placebo (one tablet a day orally).
  Interventions: Diagnostic Test: Maximal functional capacity by cardiopulmonary exercise testing; Diagnostic Test: Echocardiography; Behavioral: Evaluation of health related quality of life; Diagnostic Test: Submáximal functional capacity assesment by 6 minutes walk test; Other: Clinical evaluation

INTERVENTIONS:
Diagnostic Test: Maximal functional capacity by cardiopulmonary exercise testing — It will be done with cycle ergometer (CORTEX Metamax3B), starting with 10W of power and increasing 10W every minute. During the test, heart rate, rhythm and blood pressure will be monitored. Gas exchange data shall be evaluated every 10 seconds and the peak oxygen consumption (peak VO2) shall be considered the maximum value obtained during the last 20 seconds of exercise. The main parameters to be determined are: maximum functional capacity, peak VO2, slope of the VE/VCO2 ratio, and chronotropic incompetence variables. It will be performed by a trained cardiologist blind to study treatment at baseline and at 30 and 90 days after treatment initiation.
  Other Names: peak oxygen consumption
Diagnostic Test: Echocardiography — The following parameters will be evaluated: a)left ventricular volumes; b) left ventricular systolic function; and c)left atrial volume and E/e' ratio. It will be performed by a trained cardiologist blind to study treatment at baseline and at 30 and 90 days after treatment initiation.
  Other Names: Diastolic and Systolic function
Behavioral: Evaluation of health related quality of life — Assessment of the quality of life through the Minnesota Living with Heart Failure Questionnaire (MLHFQ), Spanish version. It will be completed at baseline and at 30 and 90 days after treatment initiation. The score of the questionnaire is 0 to 105 points.
  Other Names: Quality of life
Diagnostic Test: Submáximal functional capacity assesment by 6 minutes walk test — It will be performed in an area equipped for cardiopulmonary resuscitation. Subjects will be asked not to perform a vigorous physical exercise in the previous 2 hours. They will be allowed to have a light meal before the test. Before the test, the vital signs will be determined in a seated position after a rest of 10 minutes. Subjects will be instructed to walk at their own pace to cover as much distance as possible in 6 minutes. It will be performed by a trained nurse blind to study treatment at baseline and at 30 and 90 days after treatment initiation.
  Other Names: 6 minutes walk test
Other: Clinical evaluation — Evaluation of signs and symptoms of heart failure

SUMMARY:
This study will be a double-blind multicenter randomized study (1:1) to evaluate the effect of dapagliflozin 10 mg per day or placebo on short-term functional capacity evaluated through changes in peak oxygen consumption.

DETAILED DESCRIPTION:
This study will be a double-blind multicenter randomized study (1:1) to evaluate the effect of dapagliflozin 10 mg per day or placebo on short-term functional capacity evaluated through changes in peak oxygen consumption. This trial will include patients with stable symptomatic heart failure with reduced ejection fraction (HFrEF). Efficacy endpoints will be evaluated at 3 time points: 1) baseline (before dapagliflozin/placebo administration), 2) 30 days after randomization, and, 3) 90 days after randomization. An intermediate clinical visit will be performed one week after study initiation.

Pre-and post-treatment evaluations (at baseline, 30 and 90 days) will include clinical assessment, cardiopulmonary exercise stress test, echocardiography, 6-minute walk test (6MWT), and quality of life indicators (Minnesota Living with Heart Failure Questionnaire -MLHFQ).

The investigators postulate that dapagliflozin 10 mg/day improves short-term functional capacity of patients with symptomatic HFrEF through multifactorial mechanisms, such as diuretic effect and improvement in myocardial energetic efficiency.

ELIGIBILITY:
Inclusion Criteria:

* The participant or his legal representative is willing and able to give informed consent for participation in the study.
* Male or female, aged ≥18 years.
* Established documented diagnosis of symptomatic HF (NYHA functional class II-III), which has been present for at least 2 months.
* LVEF ≤40% documented in the last 3 months by echocardiography or cardiac magnetic resonance.
* NT-proBNP ≥600 pg/ml.
* Patients should receive background standard of care for HFrEF at judgment of the investigator.
* Estimated glomerular filtration rate (eGFR) ≥30 ml/min/1.73m2 (DMRD formula) at enrolment.

Exclusion Criteria:

* Inability to perform a valid (respiratory exchange ratio -RER- ≥1.05) baseline cardiopulmonary exercise test (CPET)
* Patients receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrolment, or previous intolerance of an SGLT2 inhibitor
* Type 1 diabetes
* Symptomatic hypotension or systolic blood pressure <95 mmHg
* Current acute decompensated HF or hospitalization due to decompensated HF <4 weeks prior to enrolment
* Myocardial infarction, unstable angina, stroke, or transient ischemic attack within 12 weeks prior to enrolment
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) or cardiac valve repair/replacement within 12 weeks prior to enrolment, or planned to undergo any of these operations after randomization
* Implantation of a cardiac resynchronization therapy (CRT) device within 12 weeks prior to enrolment or intent to implant a CRT device
* Previous cardiac transplantation or implantation of a ventricular assistance device or similar device, or implantation expected after randomization
* HF due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy, or uncorrected severe primary cardiac valve disease
* Symptomatic bradycardia or second or third-degree heart block without a pacemaker
* Severe renal dysfunction (eGFR<30 ml/min/1.73m2) or prior admission for acute renal failure in the last 4 weeks.
* Pregnant or lactating women
* Woman of childbearing age, unless they are using highly effective contraceptive methods.
* Patients with severe hepatic impairment (Child-Pugh class C).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Functional capacity | At baseline, 30 and 90 days after starting treatment with dapagliflozin or placebo.
  Changes in peak oxygen consumption (VO2) at baseline, 30 and 90 days after starting treatment with dapagliflozin or placebo. VO2 is only one measure and is expressed as milliliters of oxygen per kilogram of body weight per minute (oxygen in milliliters, weight in kilograms, and time in minutes and expressed in ml/kg/min).

SECONDARY OUTCOMES:
Left ventricular volumes | At baseline, 30 and 90 days after starting treatment with dapagliflozin or placebo.
  The following parameters will be evaluated:
  Left ventricular diastolic volume (measured in milliliters, mL) and systolic volume (measured in milliliters, mL) It will be performed by a trained cardiologist blind to study treatment at baseline and at 30 and 90 days after treatment initiation.
Left ventricular ejection fraction | At baseline, 30 and 90 days after starting treatment with dapagliflozin or placebo.
  The following parameter will be evaluated:
  Left ventricular ejection fraction (measured by simpson method and expressed in percentage, %).
  It will be performed by a trained cardiologist blind to study treatment at baseline and at 30 and 90 days after treatment initiation.
Left atrial volume | At baseline, 30 and 90 days after starting treatment with dapagliflozin or placebo.
  The following parameter will be evaluated:
  Determination of 2-dimensional derived left atrial volume (volumen measured in milliliters, mL) indexed for body surface area (body surface area expressed in square meters -m2-) and expressed in mL/m2.
  It will be performed by a trained cardiologist blind to study treatment at baseline and at 30 and 90 days after treatment initiation.
Echocardiographic parameters of diastolic function | At baseline, 30 and 90 days after starting treatment with dapagliflozin or placebo.
  The following parameter of diastolic function will be evaluated:
  - E/e' ratio: value of E velocity-expressed in cm/s- / averaged value of septal and lateral side e´velocity - expressed in cm/s- of the mitral annulus by pulsed tissue Doppler.
  It will be performed by a trained cardiologist blind to study treatment at baseline and at 30 and 90 days after treatment initiation.
Evaluation of health related quality of life by Minnesota Living with Heart Failure Questionnaire (MLHFQ) | At 30 and 90 days after starting treatment with dapagliflozin or placebo.
  Assessment of the quality of life through the Minnesota Living with Heart Failure Questionnaire (MLHFQ). It will be completed at baseline and at 30 and 90 days after treatment initiation. The score values are ranged between 0 to 105 points.
Submáximal functional capacity assesment by 6 minutes walk test | at 30 and 90 days after starting treatment with dapagliflozin or placebo.
  It will be performed in an area equipped for cardiopulmonary resuscitation. Subjects will be asked not to perform vigorous physical exercise in the previous 2 hours. They will be allowed to have a light meal before the test. Before the test, the vital signs will be determined in a seated position after a rest of 10 minutes. Subjects will be instructed to walk at their own pace to cover as much distance (measured in meters) as possible in 6 minutes. It will be performed by a trained nurse blind to study treatment at baseline and at 30 and 90 days after treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Nuñez Villota, Principal Investigator — Fundación para la Investigación del Hospital Clínico de Valencia
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nunez J, Palau P, Dominguez E, Mollar A, Nunez E, Ramon JM, Minana G, Santas E, Facila L, Gorriz JL, Sanchis J, Bayes-Genis A. Early effects of empagliflozin on exercise tolerance in patients with heart failure: A pilot study. Clin Cardiol. 2018 Apr;41(4):476-480. doi: 10.1002/clc.22899. Epub 2018 Apr 17. PMID 29663436
- [Derived] Lorenzo M, Jacobs-Cacha C, Palau P, Amiguet M, Seller J, Nunez E, Espriella R, Gorriz JL, Minana G, Sanchis J, Bayes-Genis A, Soler MJ, Packer M, Nunez J; DAPA-VO2 Investigators. Short-Term Changes in Peak VO2 After Initiation of Dapagliflozin in Heart Failure Across Iron Status. JACC Heart Fail. 2023 Nov;11(11):1611-1622. doi: 10.1016/j.jchf.2023.07.010. Epub 2023 Sep 6. PMID 37676213
- [Derived] Amiguet M, Palau P, Dominguez E, Seller J, Pinilla JMG, de la Espriella R, Minana G, Valle A, Sanchis J, Gorriz JL, Bayes-Genis A; DAPA VO2 investigators; Nunez J. Dapagliflozin and short-term changes on circulating antigen carbohydrate 125 in heart failure with reduced ejection fraction. Sci Rep. 2023 Jun 30;13(1):10591. doi: 10.1038/s41598-023-37491-5. PMID 37391470
- [Derived] Palau P, Amiguet M, Dominguez E, Sastre C, Mollar A, Seller J, Garcia Pinilla JM, Larumbe A, Valle A, Gomez Doblas JJ, de la Espriella R, Minana G, Mezcua AR, Santas E, Bodi V, Sanchis J, Pascual-Figal D, Gorriz JL, Bayes-Genis A, Nunez J; DAPA-VO2 Investigators (see Appendix). Short-term effects of dapagliflozin on maximal functional capacity in heart failure with reduced ejection fraction (DAPA-VO2 ): a randomized clinical trial. Eur J Heart Fail. 2022 Oct;24(10):1816-1826. doi: 10.1002/ejhf.2560. Epub 2022 Jun 6. PMID 35604416